CLINICAL TRIAL: NCT04148131
Title: Viscoelastic Properties of the Denervated Muscles in Children With Upper Trunk Obstetrical Brachial Plexus Palsy
Brief Title: Muscle Viscoelastic Properties In Birth Palsy
Acronym: Birth Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kıvanç Delioğlu, Principal Investigator, MSc, Hacettepe University
Other Study IDs: kıvançOBPP
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Birth Injuries; Obstetric; Injury
Keywords: Brachial Plexus; birth injury
MeSH Terms: conditions — Birth Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1, 0-5 months old: Children which is Obstetric brachial plexus palsy and 0-5 months old age have Naracas type 2 lesion.
- Group 2, 6-24 months old: Children which is Obstetric brachial plexus palsy and 6-24 months old age have Naracas type 2 lesion.
- Group 3, 25-36 months old: Children which is Obstetric brachial plexus palsy and 25-36 months old age have Naracas type 2 lesion.

SUMMARY:
The aim of study was to observe changes in denervated muscles viscoelastic properties and motor performance of OBPP children. Viscoelastic properties have a significant effect on muscle performance; however have not investigated yet in denervated muscle. Hypothesized that the viscoelastic properties of denervated muscles are different than healthy side muscles and can vary depending on the age groups. 74 patients who have C5-C6 root lesion were enrolled to the study. The patients were grouped according to their age groups: 1-5 months, 6-24 months and 25-36 months. Myoton-3 myotonometric measuring device was used to measure the viscoelastic properties (tone, elasticity and stiffness) of deltoid, biceps brachii. Active Movement Scale were used to evaluate the motor function of the muscles. There were difference in muscle viscoelastic properties depending on age group. Children aged 0-5 months showed significant difference in deltoid muscle tone (p=0.0001), stiffness (p=0.0001), biceps brachii muscle tone (p=0.0001) and stiffness (p=0.0001), when compared with other groups (denervated side was lower in values).

Therefore, it is in our opinion that in follow-up, clinical assessment of viscoelastic properties will be useful for monitoring denervated muscle; also treatment programs and purposes for OBPP should be varying according to the muscle properties.

DETAILED DESCRIPTION:
Birth lesion of the brachial plexus, generally referred as "obstetric brachial plexus palsy (OBPP)", frequently includes traction or tearing of the nerve plexus that supply motor, sensory and autonomic innervation to the arm. The extent of damage can vary depending on severity of the injuries; from single nerve root to total root lesions. Impact of OBPP can be seen as transient functional insufficiencies to lifelong total disability, depending on the injury severity. The incidence of OBPP varies between 1.3 - 1.5 per 1000 births in different countries. The most common risk factor for birth injury is shoulder dystocia. Other risk factors are macrosomia, prolonged labor, multiparity, maternal pelvic anatomy and ethnic background.Denervation after delivery leads changes in the muscle tissue due to incomplete maturation of the muscles. The muscle tissue cannot grow longitudinally and have higher connective tissue content. Additionally, muscle strength gain, and development are impaired in the denervation process due to fibrosis and fat infiltration. Many studies demonstrated alterations in histomorphological features of denervated muscles in OBPP via magnetic resonance, ultrasound imaging and gene analysis. Despite many structural alterations in muscles have been investigated; changes in the viscoelastic properties, including muscle tone (tonus), stiffness and elasticity of the muscles, during denervation and reinnervation processes have not yet been investigated in patients with OBPP. The aim of our study was to observe changes in denervated muscles viscoelastic properties and motor performance of OBPP children. Viscoelastic properties have a significant effect on muscle performance; however have not investigated yet in denervated muscle. Hypothesized that the viscoelastic properties of denervated muscles are different than healthy side muscles and can vary depending on the age groups. 74 patients who have C5-C6 root lesion were enrolled to the study. The patients were grouped according to their age groups: 1-5 months, 6-24 months and 25-36 months. Myoton-3 myotonometric measuring device was used to measure the viscoelastic properties (tone, elasticity and stiffness) of deltoid, biceps brachii. Active Movement Scale were used to evaluate the motor function of the muscles. We found different muscle viscoelastic properties depending on age group. Children aged 0-5 months showed significant difference in deltoid muscle tone (p=0.0001), stiffness (p=0.0001), biceps brachii muscle tone (p=0.0001) and stiffness (p=0.0001), when compared with other groups (denervated side was lower in values).Therefore, it is in our opinion that in follow-up, clinical assessment of viscoelastic properties will be useful for monitoring denervated muscle; also treatment programs and purposes for OBPP should be varying according to the muscle properties.

ELIGIBILITY:
Inclusion Criteria:

* Our inclusion criteria were; having only C5-C6 root injury, being classified as Narakas type 2,
* being treated with conventional physiotherapy and routinely followed up by our clinic since birth.

Exclusion Criteria:

* Our exclusion criteria were having a root injury other than C5-C6,
* having a history of orthopaedic or neurologic surgery,
* having low birth weight or premature birth history,
* having a systemic, genetic or neuromuscular disease.

Max Age: 36 Months | Sex: All
Age Groups: Child
Study Population: * The Population have Obstetric Brachial Plexus Palsy
  * Seventy-four (25 boys, 49 girls) children aged between 1-36 months (15.12±10.58) with Narakas type 2 injury (C5-C6 upper trunk involvement) were enrolled to the study
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Myotone-3, Viscoelastic Properties Measurement | a day (single measurement)
  Viscoelastic properties of deltoid and biceps brachii muscles in both denervated and healthy sides were analyzed with using Myoton-3 device, which is a reliable handhold device for measuring viscoelastic properties of muscles by recording the damped mechanical oscillations; and provides objective, painless and noninvasive way to measure quantitative value of the muscle tone, stiffness and elasticity, invented at the University of Tartu in Estonia (Müomeetria AS, Estonia, EU) (ICC: 0,80-0,93).

SECONDARY OUTCOMES:
Active Movement Scale | a day (single measurement)
  The Active Movement Scale (AMS) was developed, specifically for children with OBPP, to investigate motor performance of denervated upper extremity and to evaluate 15 motions in upper extremity. The scoring system uses a 7-point scale for movement, based on the percentage of active movement observed considering full range of motion for each joint. 0-4 points are given for movement of the joint in the gravity minimized position. Points 5-7 are given based on performing activities against gravity.

IPD SHARING:
Plan to Share IPD: No